CLINICAL TRIAL: NCT06105658
Title: A Clinical Study to Evaluate the Safety and Efficacy of Unrelated Umbilical Cord Blood Microtransplantation in Patients With Acute Myelocytic Leukemia
Brief Title: Safety and Efficacy of Unrelated Umbilical Cord Blood Microtransplantation in Patients With AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Principal Investigator, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCB-MST&AML
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy+unrelated umbilical cord blood microtransplantation (Experimental): Intermittent infusion of HLA mismatched or incompletely matched granulocyte colony-stimulating factor (G-CSF) mobilized peripheral blood stem cells (G-PBSC) during routine chemotherapy without the use of immunosuppressants, abbreviated as "microtransplantation".
  Interventions: Biological: Unrelated umbilical cord blood; Drug: Venetoclax; Drug: Decetabine; Drug: Azacitidine

INTERVENTIONS:
Biological: Unrelated umbilical cord blood — The requirements of unrelated umbilical cord blood: recipient-donor HLA match is 0-3/10, same blood type.
Drug: Venetoclax — Patients will be treated with Venetoclax (100 mg on day 1, 200 mg on day 2 and 400 mg on days 3 to 21)
Drug: Decetabine — Patients will be treated with Decetabine (20mg/m^2/d on days 1 to 5) or Azacitidine (75mg/m^2/d on days 1 to 7)
Drug: Azacitidine — Patients will be treated with Decetabine (20mg/m^2/d on days 1 to 5) or Azacitidine (75mg/m^2/d on days 1 to 7)

SUMMARY:
This study aimed to evaluate the safety and efficacy of unrelated umbilical cord blood microtransplantation in the treatment of AML patients by observing the factors related to the efficacy and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with AML through bone marrow morphology, histochemistry, immunophenotyping, pathological testing, etc. Besides, patients should meet the following conditions:

   Patients aged 60-80 who newly diagnosed AML with WHO criteria and have not received prior treatment for acute leukemia (hydroxyurea or pre-chemotherapy is allowed for patients with high leukocyte).

   Patients aged 14-60 who do not meet the indications for hematopoietic stem cell transplantation;
2. Gender and race are not limited;
3. Karnofsky score ≥ 60%, Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
4. Expected survival time ≥ 3 months;
5. The examination results meet the following requirements:

   ALT and AST ≤ 3 × Upper limit of normal value (ULN); Total bilirubin ≤ 3 × ULN; Creatinine ≤ 2 × ULN or creatinine clearance rate ≥ 40mL/min; The left ventricular ejection fraction (LVEF) measured by echocardiography or multigated acquisition (MUGA) scanning is within the normal range (>50%);
6. The recipient and selected donor should be 0-3/10 HLA-matched with same blood type;
7. Patients who voluntarily participate in this clinical study and have signed an informed consent.

Exclusion Criteria:

1. Patients who have suffered from malignant tumors;
2. Patients have suffered from hematopoietic failure after chemotherapy, and have undergone ineffective blood transfusion with unknown cause;
3. Patients who have undergone Class II or above surgery within 4 weeks prior to enrollment;
4. Suffering from life-threatening diseases other than AML;
5. Allergic to the drugs in the research;
6. Patient with severe cardiac insufficiency, including uncontrolled or symptomatic arrhythmia, congestive heart failure, myocardial infarction within 6 months, or any grade 3 (moderate) or grade 4 (severe) heart disease;
7. Patients with test positive for HIV, HCV or HBV;
8. Stroke or intracranial hemorrhage occurred within 6 months prior to enrollment;
9. Warfarin or vitamin K antagonists (such as phenprocoumarin) is necessary for anticoagulation;
10. Patients with mental illnesses or cognitive impairments;
11. Patients have participated within the month prior to enrollment or patients are currently participating in other clinical trials;
12. There are other conditions that the investigators consider inappropriate for inclusion.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 28±7days
  CR rate is defined as the percentage of patients who met the following conditions:
  Myelogram: naïve cells less than 5% (at least 200 nucleated cells); Hemogram: absolute neutrophil count > 1.0×10^9/L, platelet count > 100×10^9/L; Clinical diagnosis: no symptoms and signs caused by leukemia infiltration, and patients do not rely on blood transfusion.
Hematopoietic recovery time | 28±7days
  The time of absolute neutrophil count>0.5×10^9/L and platelet count >30×10^9/L for 3 consecutive days.

SECONDARY OUTCOMES:
Time to Progression（TTP） | 1 year
  Time from enrollment to objective progression of disease
Disease Free Survival（DFS） | 1 year
  From CR to recurrence or death or to the date of last follow-up
Overall Survival（OS） | 1 year
  From the beginning of treatment to death or to the date of last follow-up
Early mortality rate | 3 months
  Death within the first 3 months of induction therapy

OTHER OUTCOMES:
Changes in lymphocyte subsets (NK cells, T cells) before and after treatment | At the time of enrollment and at 1 month
  The concentration of lymphocyte subsets in peripheral blood can be detected by flow cytometry
Correlation between human leukocyte antigen (HLA) matching and the concentration of lymphocyte subsets | HLA typing and matching will be assessed at the time of enrollment, and the concentration of lymphocyte subsets in peripheral blood will be detected at the time of enrollment and at 1 month
  HLA typing and matching can be assessed by sequence based genotyping (PCR-SBT), and the concentration of lymphocyte subsets in peripheral blood can be detected by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, MD, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China